CLINICAL TRIAL: NCT04453267
Title: DNA Repair in Patients With Stable Angina.
Acronym: DECODE II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CAR0566
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis; DNA Damage; DNA Repair Abnormality
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stored samples of isolated T-Cells and Monocytes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Arm.: Consecutive patients undergoing elective percutaneous coronary intervention (PCI) or isolated coronary artery bypass grafting (CABG) for symptomatic stable angina (SA) despite optimal medical therapy at the University Hospital Southampton NHS Foundation Trust will be prospectively enrolled (n=86).
  No interventions administered. 40ml of whole blood in EDTA vials to be taken for cellular separation and analysis.
- Age and gender matched controls: Age and gender-matched patients being investigated for chest pain with unobstructed coronary arteries, defined as coronary stenosis ≤ 30% in any major epicardial vessel on CT or invasive coronary angiography, will also be recruited as controls (n=86).
  40ml of whole blood in EDTA vials to be taken for cellular separation and analysis.

SUMMARY:
Markers of DNA damage and repair are present in both atherosclerotic plaques and peripheral blood mononuclear cells of patients with coronary artery disease. A positive correlation has been observed between the level of DNA damage and the severity of atherosclerotic lesions, as well as atherogenic risk factors such as smoking, hypertension and hyperlipidaemia. A number of in-vitro studies have implicated defective DNA repair in the development and progression of atherosclerotic lesions. In mouse models of atherosclerosis, the DNA repair signalling cascade has been shown to be amenable to pharmacological intervention and overexpression of specific repair proteins attenuate the development of atherosclerotic plaques. However, data regarding the role of DNA repair in the pathogenesis of atherosclerosis in humans are lacking. We have preliminary data indicating reduced DNA repair activity in patients with stable angina. This study will determine the molecular basis and the biological consequences of this observation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to provide written informed consent

Exclusion Criteria:

* Age ≥ 80 years
* Inability to provide written informed consent
* Presentation with an acute coronary syndrome
* Severe valvular heart disease
* Hypertrophic cardiomyopathy
* Left ventricular ejection fraction ≤ 35%
* Prior coronary revascularisation (surgical or percutaneous)
* Diabetes Mellitus
* Clinical evidence of peripheral vascular disease
* Prior history of cerebrovascular disease
* Malignancy
* Active inflammatory disorders (e.g. rheumatoid arthritis/connective tissue disorder)
* Renal impairment eGFR <60ml/min/1.73m2
* Anaemia (Hb <100g/dL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an assessment of thier coronary anatomy either by computerised tomography coronary angiogram or invasive coroanry angiogram at a large university teaching hospital performed as part of thier routine care.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Association between monocytes exhibiting reduced base excision repair and/or double strand break repair activity in patients with stable angina as compared to patients without coronary artery disease. | Blood will be collected at the time of hospital admission for index procedure. No follow-up of patients will be required.
  This will be assessed using real-time polymerase chain reaction, western blotting and proteosomal degradation assay.
Reduced DNA repair activity is associated with impaired response to oxidative stress in human monocytes in patients with stable angina in comparison to an age and gender matched control. | Blood will be collected at the time of hospital admission for index procedure. No follow-up of patients will be required.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mahmoudi, MD,PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No